CLINICAL TRIAL: NCT03020394
Title: Comparison of High Flow Nasal Cannula, Noninvasive Positive Ventilation (NPPV) and Invasive Positive Ventilation (IPPV) in Severe Chronic Obstructive Pulmonary Disease Exacerbation (AECOPD)
Brief Title: Respiratory Support in Severe Chronic Obstructive Pulmonary Disease Exacerbation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Qingyuan Zhan, Head of Pulmonary and Critical care medicine ward 4, China-Japan Friendship Hospital
Other Study IDs: 2016YFC1304304-3
Record Dates: First submitted 2017-01-09; First posted 2017-01-13 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: COPD Exacerbation
Keywords: COPD Exacerbation; Noninvasive Positive Ventilation; Invasive Positive Ventilation; severe; High flow nasal cannula
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Noninvasive ventilation: Noninvasive positive pressure ventilation is achieved by Philips Respironics V60/Vision ventilator. Choose bilevel positive airway pressure mode, and adjust the fraction of inspire oxygen(FiO2) or oxygen flow rate to maintain patient's oxygen saturation(SpO2) between 88% to 92%. Parameter adjustment and weaning of NPPV follow the protocols used before.
- Invasive ventilation: Intubated immediately and connected to the ventilator. Parameter adjustment and weaning of IPPV follow the protocols used before.
- High flow nasal cannula: High flow nasal cannula of different models (large, medium and small) are selected depending on the size and comfort of the patient's nostrils. Adjusting the oxygen flow rate (O2 Flow) maintains the patient's SpO2 88% to 92%. The flow was initially adjusted to 25 L/min and the flow was gradually adjusted to the patient's maximum tolerance. The inspiratory gas temperature (31 to 37 °C) was set to the patient's maximum tolerance level. If the patient's condition deteriorates and the tracheal intubation standard is met , the patient is recommended to undergo invasive ventilation treatment, but the choice of the final respiratory support method should be decided by the attending physician, patient and family.

SUMMARY:
Preliminary studies have shown that NPPV can avoid tracheal intubation in 40% to 60% patients who have severe exacerbation of COPD. Recently, large-scale comparative effectiveness research (CER) also found that compared with invasive ventilation, NPPV can reduce mortality rates. But there's no high-quality clinical studies which can confirm this. Therefore, investigators believe that NPPV can avoid intubation in patients with severe exacerbation of COPD in ICU with perfect monitoring conditions and reasonable human resource allocation, in order to reduce IMV-related complications and improve patients' outcomes.

DETAILED DESCRIPTION:
In part of the patients who were AECOPD with pH <7.25 , preliminary studies have shown that NPPV can avoid tracheal intubation in 40% to 60% patients, and also reduce the incidence of VAP. Recently, large-scale comparative effectiveness research (CER) also found that compared with invasive ventilation, NPPV can reduce mortality rates. At present, there's no high-quality clinical studies which can confirm this, and clinical guidelines do not have a recommendation on the use of NPPV in these patients. Therefore, investigators believe that NPPV can avoid intubation in patients with severe exacerbation of COPD in ICU with perfect monitoring conditions and reasonable human resource allocation, as well as the progress of medical technology in NPPV in recent years, in order to reduce IMV-related complications and improve patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD;

Exclusion Criteria:

* refuse to engage in the study;
* have been included in other study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute exacerbation of chronic obstructive pulmonary disease in medical ICU.
Sampling Method: Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of ventilator-associated pneumonia (VAP) | 90days
The all cause mortality of ICU and hospitalization | 90 days

SECONDARY OUTCOMES:
The length of stay of ICU and hospitalization | 90 days
The length of stay of mechanical ventilation | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Qingyuan Zhan, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No